CLINICAL TRIAL: NCT01981018
Title: Mood Action Psychology Programme (MAPP): a Case Series Investigation of Brief Imagery-focused Cognitive Therapy (imCT) for Bipolar Disorder.
Brief Title: MAPP: Imagery-focused Therapy for Bipolar Disorder
Acronym: MAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council Cognition and Brain Sciences Unit (Other Government)
Collaborators: Cambridgeshire and Peterborough NHS Foundation Trust (Other); Oxford Health NHS Foundation Trust (Other Government); University of Cambridge (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAPP_0174
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Bipolar Disorder
Keywords: Mental imagery, CBT, anxiety, mood instability
MeSH Terms: conditions — Bipolar Disorder; Color Vision Defects; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imagery-focused Cognitive Therapy (Experimental): 10 sessions of imagery-focused Cognitive Therapy delivered approximately weekly by two co-therapists, divided in 4 assessment, 4 treatment and 4 consolidation sessions; additional 2 "blip" management sessions during therapy and 3 "blip" management and booster session during follow up can be delivered if necessary.
  Interventions: Other: Imagery-focused Cognitive Therapy (ImCT - psychotherapy based on CBT principles)

INTERVENTIONS:
Other: Imagery-focused Cognitive Therapy (ImCT - psychotherapy based on CBT principles) — ImCT Therapy is carried out by a team of 2 co-therapists and comprises of:
  * Mapping: Therapists and patient collaboratively map out difficulties and pinpoint a treatment focus, with regards to imagery symptoms and anxiety co-morbidity that impact on bipolar mood instability. This leads to an individualised formulation of the patient's current problem.
  * Target: Follows the rationale, timing and objectives identified collaboratively in Mapping. It is structured around imagery-based techniques, such as imagery rescripting, which are used to address problematic imagery, to promote management of mood and boost self-care. This results into the acquisition of imagery-based mood- and anxiety-regulating strategies to be integrated into the patient's already existing coping strategies.
  * Consolidation: Consist of fine tuning the strategies devised during Target based on experience gained after testing them out in real life situations and includes a "video blue print.

SUMMARY:
Bipolar Disorder (BD) (previously known as "manic depression") is a severe mental health illness affecting at least 1% of the population and with annual NHS cost estimated at £342 million. It is characterised by alternating episodes of acute mood swings: depression and "mania" (mood elation). BD also comes with less severe mood swings we call "mood instability", and ongoing high levels of anxiety that impair well-being even during periods between the acute mood breakdowns. Anxiety and mood instability are associated with worse outcome of the disorder.

All these symptoms can be accompanied by the presence of troublesome mental images (e.g. seeing a memory in the mind's eye) such as intrusive "flashbacks" of negative past events. Recent studies suggest that individuals with BD experience more vivid, compelling and upsetting mental images compared to other patient groups and this could contribute to their clinical difficulties.

Cognitive Behavioural Therapy (CBT) is a well established and successful psychological therapy used in the National Health Service (NHS), UK but as yet with limited efficacy in BD. Targeting mental imagery has long been part of general CBT. In particular, imagery-based treatment techniques have proved successful in anxiety disorders, but have not been brought to CBT for Bipolar Disorder yet.

Our study Mood Action Psychology Programme (MAPP) investigates the delivery of a brief imagery-focused cognitive therapy (imCT) intervention to people with BD, studying a series of patients in detail one by one a "case series"). We offer a structured and individualised psychological treatment in line with the aims of NHS guidelines. The imCT protocol has been successfully delivered and audited in our psychological service in Oxford (OxMAPP). The proposed MAPP study aims to formally assess for the first time the effectiveness of imCT. In particular we hypothesise that imCT via the Mood Action Psychology Programme (MAPP) will result in (i) reduced levels of anxiety and (ii) reduced levels of low mood after treatment compared to baseline (both measured over 4 weeks) in individuals with BD.

Overall, this works aims to contribute to improved psychological treatment for BD.

DETAILED DESCRIPTION:
Mood Action Psychology Programme (MAPP) is a study that investigates the delivery of an imagery-focused cognitive therapy (imCT) intervention to people with Bipolar Disorder (BD) via a single case series (N = 15) design. MAPP offers patients a structured and individualised psychological treatment (imCT) for BD inline with the aims of the National Institute for Clinical Excellence, UK guidelines (NICE, 2006) and as already developed and audited in the OxMAPP psychological service that was run within the Professorial Mood Disorders clinic at the Warneford Hospital, Oxford. In addition MAPP aims to improve the understanding of psychological therapy by formally assessing the effectiveness of imCT in reducing anxiety and low mood symptoms. Secondary aims are to test the hypothesis that reductions in anxiety and low mood levels are mediated by changes in problematic imagery phenomena, and investigating the impact of imCT on interepisodic mood instability, coping skills and general functioning of patients with BD. The short term (i.e. at 6 month follow up) effect on preventing relapses of (hypo)manic and depressive episodes is also evaluated. The rationale for this approach derives from current evidence of (i) the uncertain efficacy in BD of traditional CBT relying exclusively on verbal thought modification approaches (Scott et al., 2006), (ii) the presence of dysfunctional mental imagery in BD patients (Bonsall et al., 2012; Hales et al., 2011; Ivins et al., under review) alongside high rates of anxiety comorbidity (Simon et al., 2004) and (iii) the success of imagery-based treatment techniques in anxiety disorders such as PTSD and social phobia (Ehlers & Clark, 2008). A case-series approach allows flexible and feasible but robust testing of the novel imCT treatment protocol with the aim of optimising it for further investigation in future randomised controlled clinical trials.

MAPP provides structured individualised treatment, which includes an extended mapping (i.e. assessment) phase for patients with BD based on cognitive behavioural principles. Where appropriate, MAPP offers a brief cognitive therapy intervention drawing on mental imagery (imCT). It includes a focus on addressing anxiety symptoms that are often present and problematic in BD. The patients and clinician jointly identify an agreed treatment target (e.g. trauma memories, social anxiety, intrusive imagery) which is hypothesised to have impact on the mood stability of patients. The agreed treatment target is one which is judged to be tractable and amenable to change in a brief intervention using imagery focused techniques.

Participation in the MAPP study is suitable for outpatients with a diagnosis of BD who would like to gain a better understanding of their symptoms, are interested in adding a psychological approach to their mood management, and are happy to take part in clinical research. The programme involves weekly symptom monitoring, as well as committing to weekly therapy sessions (10 sessions), and is suitable for patients who are agreeable to both of these. Treatment is offered to patients who comply with the daily mood monitoring active run in phase. Referrals of young patients (18-25 years old) are encouraged, given evidence that psychological treatment might be more effective at the onset of BD, in particular when targeting anxiety and mood instability. Within MAPP, psychological treatment is delivered by a team of therapists. The therapists are clinical psychologists and psychiatrists with specific imCT training. Typically two co-therapists are present in each session, one of which can attend the session also via Skype. MAPP is integrated in psychiatric secondary care within two NHS trusts, the Cambridge and Peterborough Foundation NHS Trust and the Oxford Health NHS Foundation Trust. In both NHS trusts imCT is given alongside psychiatric medication as usual. Patients enrolled in the study maintain their ongoing contact with other core clinical services.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 - 65 years old
* Have adequate English language ability to permit the assessment and experimental measures to be completed
* Have diagnosis of Bipolar Disorder (I or II or NOS) according to Diagnostic and Statistical Manual IV-TR (DSM-IV) criteria (American Psychiatric Association, 2000) as indicated by the Structured Clinical Interview for DSM-IV (SCID) (First, Spitzer, M., & Williams, 2002)
* Are willing to complete daily/weekly mood and anxiety monitoring throughout the duration of the study
* Successfully complete daily monitoring in the 4 weeks active run-in phase
* Are willing to have regular treatment reports and letters sent to their GP and other relevant clinicians
* Can commit to attending 10 consecutive weekly sessions, including questionnaires completion, and follow up period as required by the study
* Are residents within geographical areas covered by the NHS trusts where treatment is delivered

Exclusion Criteria:

* Do not have diagnosis of Bipolar Disorder (I or II or NOS) according to Diagnostic and Statistical Manual IV-TR (DSM-IV) (American Psychiatric Association, 2000) criteria as indicated by the Structured Clinical Interview for DSM-IV (First et al., 2002)
* Learning difficulties, organic brain disease, severe neurological impairment
* Current severe substance or alcohol misuse (clinicians assessment)
* Current manic episode as diagnosed by DSM-IV criteria (American Psychiatric Association, 2000) indicated by the SCID (First et al., 2002)
* Current active psychotic symptoms
* Presence of active suicidal risk as indicated by a score of 2 or more on item 12 of the QIDS (Rush et al., 2003) (i.e. frequent thoughts and/or plans to end their life) confirmed by convergent clinical opinion
* Unwilling to engage actively in treatment or to use an imagery-focussed approach for treatment
* Taking part in concurrent treatment studies investigating pharmacological or psychological treatment for BD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Anxiety and depression scores change | 4 weeks
  To assess the primary endpoint in the study, i.e the change in scores on measures of (i) Beck Anxiety Inventory (BAI) (Beck & Steer, 1993) (ii) Quick Inventory of Depressive Symptoms (QIDS) (Rush et al., 2003) after treatment, pooled scores from aggregated time points over 4 weeks after treatment compared to aggregated time points over baseline changes anxiety (BAI) and low mood (QIDS) are used. This method is advised given that traditional self-report mood ratings over a single time point are scarcely representative of mood variability in BD. For this scope the following assessments are repeated weekly for all study duration:
  * Quick Inventory of Depressive Symptomatology, Self-Report (QIDS) (Rush et al., 2003)
  * Beck Anxiety Inventory (BAI) (Beck & Steer, 1993)

SECONDARY OUTCOMES:
Changes in Imagery Characteristics | 4 weeks
  Imagery characteristics are recorded in order to test if reductions in anxiety and low mood levels over 4 weeks after treatment compared to baseline (i.e. the primary objective) are mediated by reductions in levels of problematic imagery during treatment.
  This is assessed from recording changes in Visual Analogue Scales of Imagery Characteristics (VAS Imagery) combined ratings pooled from aggregated time points during treatment. Visual Analogue Scales (VAS Imagery) have been tailored to BD population rating on a scale 0-9, for example such as: "How real / vivid / absorbing / preoccupying / compelling have your image(s) been over the past week'"; "To which extent could you understand the role that the image(s) play in your mood instability?"; "To which extent could you find positive / helpful way of using the image(s)?", in line with Brewin (Brewin et al., 2009) and clinical audit results from the OxMAPP clinical psychology service for BD.
Anxiety and depression change maintenance at follow up | 12 and 24 weeks
  Change in scores on measures of (i) BAI (anxiety scale) (ii) QIDS (depression scale) will be pooled from aggregated time points over 12 and 24 weeks during follow up and compared to aggregated time points over baseline.
Mood instability | 4 weeks and 24 weeks
  Change in mood instability will be calculated as the time series profile of daily mood and anxiety ratings on the QIDS-m scale over 4 weeks, prior and after treatment based on work with Bonsall (Bonsall et al., 2012); convergent change on the self-report proxy measures of mood instability Affective Lability Scale - short version (ALS-18) (Oliver & Simons, 2004) and Internal States Scale (ISS) (Bauer, Crits-Christoph, et al., 1991) will be collected at 4, 12, and 24 week follow up.
Depression and mania relapse rate and duration | 24 weeks
  Reductions in (i) the number of relapses comparing 24 weeks prior to treatment start to 24 weeks following treatment completion: a relapse is counted as a time when a patient has experienced a depressive, (hypo)manic or mixed episode according to Diagnostic and Statistical Manual IV, DSM IV diagnostic criteria counted on the Structured Clinical Interview for DSM IV (SCID); and (ii) the duration of relapses retrospectively assessed via the SCID.
Anxiety comorbidity | 24 weeks
  Reduction of number of anxiety disorders (categorised according to DSM-IV criteria) present on SCID items F1-24, F66, F67, F25-38, F40-64, F68, from baseline to 4, 12 and 24 weeks after treatment.
Medication compliance | 24 weeks
  Change in scores on the Medication Compliance Questionnaire (Lam et al., 2003) after treatment and at 4, 12 and 24 week follow up compared to baseline.
General functioning and coping | 24 weeks
  Change in scores on the Longitudinal Interval Follow up Evaluation - Range of Impaired Functioning Tool (LIFE-RIFT) (Leon et al., 2000; Leon et al., 1999) functioning scale after treatment and at 4, 12 and 24 week follow up compared to baseline; change in scores of the "Mental Imagery and Coping with Bipolar Disorder Questionnaire" after treatment and at 4, 12 and 24 week follow up compared to baseline.
Suicidality | 24 weeks
  Change in ratings of items related to suicidality on the QIDS and on the Beck Hopelessness Scale (BHS) (Beck & Steer, 1998) after treatment and at 4, 12 and 24 week follow up compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Emily A Holmes, PhD, Principal Investigator — Medical Research Council Cognition and Brain Sciences Unit
Locations (4):
- United Kingdom (4):
  - MRC Cognition and Brain Sciences Unit, Cambridge
  - Cambridge and Peterborough NHS Foundation Trust, Cambridge
  - University of Oxford, Department of Psychiatry, Oxford
  - Oxford Health NHS Foundation Trust, Oxford

REFERENCES:
- [Background] Holmes EA, Deeprose C, Fairburn CG, Wallace-Hadrill SM, Bonsall MB, Geddes JR, Goodwin GM. Mood stability versus mood instability in bipolar disorder: a possible role for emotional mental imagery. Behav Res Ther. 2011 Oct;49(10):707-13. doi: 10.1016/j.brat.2011.06.008. Epub 2011 Jul 5. PMID 21798515
- [Background] Bonsall MB, Wallace-Hadrill SM, Geddes JR, Goodwin GM, Holmes EA. Nonlinear time-series approaches in characterizing mood stability and mood instability in bipolar disorder. Proc Biol Sci. 2012 Mar 7;279(1730):916-24. doi: 10.1098/rspb.2011.1246. Epub 2011 Aug 17. PMID 21849316
- [Background] Holmes EA, Geddes JR, Colom F, Goodwin GM. Mental imagery as an emotional amplifier: application to bipolar disorder. Behav Res Ther. 2008 Dec;46(12):1251-8. doi: 10.1016/j.brat.2008.09.005. Epub 2008 Oct 8. PMID 18990364
- [Derived] Holmes EA, Bonsall MB, Hales SA, Mitchell H, Renner F, Blackwell SE, Watson P, Goodwin GM, Di Simplicio M. Applications of time-series analysis to mood fluctuations in bipolar disorder to promote treatment innovation: a case series. Transl Psychiatry. 2016 Jan 26;6(1):e720. doi: 10.1038/tp.2015.207. PMID 26812041
- See also: Mood monitoring website used for the study - password protected access — https://webmapp.mrc-cbu.cam.ac.uk/